CLINICAL TRIAL: NCT04458883
Title: The Next Leap in Cardiac Magnetic Resonance Imaging:Cycling the Field The TITAN Study
Brief Title: The Next Leap in Cardiac Magnetic Resonance Imaging:Cycling the Field
Acronym: TITAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2-010-20
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: The main aim of the study is to build and test a cardiac-specific coil purposely assembled in house to suit the FFC-MRI whole-body prototype and to test if it could be used for clinical cardiac scans in human subject populations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myocardial Infarction Group (Experimental): Patients diagnosed with a myocardial infarction
  Interventions: Procedure: Cardiac Magnetic Resonance Imaging; Procedure: Fast Field Cycling - Magnetic Resonance Imaging
- Healthy Volunteers (Experimental): Healthy Volunteers
  Interventions: Procedure: Cardiac Magnetic Resonance Imaging; Procedure: Fast Field Cycling - Magnetic Resonance Imaging; Procedure: Electrocardiogram; Procedure: Echocardiogram

INTERVENTIONS:
Procedure: Cardiac Magnetic Resonance Imaging — Cardiac Magnetic Resonance Imaging - Cardiac Scan
Procedure: Fast Field Cycling - Magnetic Resonance Imaging — Fast Field Cycling - Magnetic Resonance Imaging Cardiac Scan
Procedure: Electrocardiogram — Electrocardiogram
  Other Names: ECG
  Arms: Healthy Volunteers
Procedure: Echocardiogram — Echocardiogram
  Arms: Healthy Volunteers

SUMMARY:
The main aim of the study is to build and test a cardiac-specific coil purposely assembled in house to suit the FFC-MRI whole-body prototype and to test if it could be used for clinical cardiac scans in human subject populations.

DETAILED DESCRIPTION:
Aberdeen scientists are at the forefront of a new type of magnetic resonance imaging (MRI), having built in-house the only two available prototypes of Fast Field-Cycling MRI in the world - and these already have clinical imaging capabilities. Fast Field-Cycling MRI switches rapidly over a range of field strengths (0.2 T to 200 µT), providing a T1 dispersion curve. This information is invisible to fixed-field scanners and uncovers unique knowledge about motion and interaction between component molecules within a tissue (i.e. water/fat/proteins). In this application the investigators wish to use their in-house expertise further to extend the capability of our Fast Field-Cycling MRI to perform cardiac imaging by building the first-ever cardiac Fast Field-Cycling MRI coil and develop cardiac pulse sequences with ECG gating. The investigators will aim to establish the normalcy of T1 dispersion curves for left ventricular myocardium in healthy volunteers, and further on to distinguish the characteristics of post-myocardial infarction scar T1 dispersion curves.

ELIGIBILITY:
Inclusion Criteria:

* Participant who is willing and able to give informed consent for participation in the study
* Healthy volunteers willing to give informed consent for participation in the study
* Patients diagnosed with a previous myocardial infarction

Exclusion Criteria:

* Unwillingness to participate
* Claustrophobia
* Contraindication to MRI scanning such as implantable cardiac devices
* Participants who have had a previous myocardial infarction in the past of which they may not be aware and this is discovered whilst being scanned on the 3T MRI scanner, or who may have any other cardiology condition that they were previously unaware will not be included in the healthy control group, even if they present themselves to us as "healthy" at the time of the study visit
* Pregnancy
* Body habitus that may preclude comfortable positioning of the volunteer in either of the MRI scanners (>50cm in diameter)
* Participants with abnormal kidney function that will preclude them from receiving a contrast agent

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Magnetic Resonance Imaging | At baseline
  Cardiac Magnetic Resonance Imaging - Cardiac Scan to assess cardiac function and T1 dispersion curves
Fast Field Cycling Magnetic Resonance Imaging | At baseline
  Fast Field Cycling Magnetic Resonance Imaging - Cardiac Scan to assess cardiac function and T1 dispersion curves

CONTACTS AND LOCATIONS:
Overall Officials: Dana Dawson, DPhil, Principal Investigator — University of Aberdeen
Locations (2):
- United Kingdom (2):
  - Cardiovascular Research Facility, Aberdeen, Aberdeenshire
  - University of Aberdeen and NHS Grampian, Aberdeen, Aberdeenshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Broche LM, Ross PJ, Pine KJ, Lurie DJ. Rapid multi-field T(1) estimation algorithm for Fast Field-Cycling MRI. J Magn Reson. 2014 Jan;238:44-51. doi: 10.1016/j.jmr.2013.10.010. Epub 2013 Oct 31. PMID 24309067
- [Background] Kimmich R, Nusser W, Winter F. In vivo NMR field-cycling relaxation spectroscopy reveals 14N1H relaxation sinks in the backbones of proteins. Phys Med Biol. 1984 May;29(5):593-6. doi: 10.1088/0031-9155/29/5/011. No abstract available. PMID 6739544
- [Background] Broche LM, Ismail SR, Booth NA, Lurie DJ. Measurement of fibrin concentration by fast field-cycling NMR. Magn Reson Med. 2012 May;67(5):1453-7. doi: 10.1002/mrm.23117. Epub 2011 Oct 24. PMID 22025420
- [Background] Broche LM, Ashcroft GP, Lurie DJ. Detection of osteoarthritis in knee and hip joints by fast field-cycling NMR. Magn Reson Med. 2012 Aug;68(2):358-62. doi: 10.1002/mrm.23266. Epub 2011 Dec 12. PMID 22161576
- [Background] Scally C, Abbas H, Ahearn T, Srinivasan J, Mezincescu A, Rudd A, Spath N, Yucel-Finn A, Yuecel R, Oldroyd K, Dospinescu C, Horgan G, Broadhurst P, Henning A, Newby DE, Semple S, Wilson HM, Dawson DK. Myocardial and Systemic Inflammation in Acute Stress-Induced (Takotsubo) Cardiomyopathy. Circulation. 2019 Mar 26;139(13):1581-1592. doi: 10.1161/CIRCULATIONAHA.118.037975. PMID 30586731
- [Background] Antonopoulos AS, Sanna F, Sabharwal N, Thomas S, Oikonomou EK, Herdman L, Margaritis M, Shirodaria C, Kampoli AM, Akoumianakis I, Petrou M, Sayeed R, Krasopoulos G, Psarros C, Ciccone P, Brophy CM, Digby J, Kelion A, Uberoi R, Anthony S, Alexopoulos N, Tousoulis D, Achenbach S, Neubauer S, Channon KM, Antoniades C. Detecting human coronary inflammation by imaging perivascular fat. Sci Transl Med. 2017 Jul 12;9(398):eaal2658. doi: 10.1126/scitranslmed.aal2658. PMID 28701474